CLINICAL TRIAL: NCT00120601
Title: The Role of Pharmacotherapy in Prevention of Relapse in Alcohol Dependence
Brief Title: Trial for the Treatment of Alcohol Dependence
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sydney (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Sydney South West Area Health Service (Other Government); South Eastern Area Health Service (Other); Wentworth Area Health Services (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X99-0277; 211177
Record Dates: First submitted 2005-07-11; First posted 2005-07-18 (Estimated); Last update posted 2005-07-18 (Estimated); Status verified 2005-06

CONDITIONS: Alcoholism
Keywords: treatment; alcohol; dependence; medication
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; Acamprosate

INTERVENTIONS:
Drug: Naltrexone
Drug: Acamprosate

SUMMARY:
The purpose of this study is to compare the effectiveness of two anti-craving medications, naltrexone versus acamprosate, in the treatment of alcohol dependence.

DETAILED DESCRIPTION:
The physical, psychological and social consequences of alcohol abuse remain a critical health problem. Every year in Australia, excessive consumption is responsible for 3,000 - 6,000 deaths and costs the community $6 billion. Approximately 15% of Australians abuse alcohol and 5% of men and 3% of women are alcohol dependent (addicted to alcohol). Better treatment for alcohol dependence is urgently needed. Treatment for alcohol dependence remains unsatisfactory. Most treatments lead to abstinence in only 1 out of 3 cases, and approximately 50% of these will relapse within 3 months of completing treatment. Two drugs (naltrexone and acamprosate) appear to interfere with the effects of alcohol on the brain that promote addiction. There is evidence that both drugs are beneficial in the treatment of alcohol dependence and both are now available in Australia. At present, no data have been reported comparing the effectiveness of these two drugs. The proposed project will compare naltrexone and acamprosate in a large, carefully performed, study. The study will help determine which subjects are likely to benefit from one or the other of these agents.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependence according to the ICD10 criteria, with alcohol as the subject's drug of choice
* Ages 18-65
* Adequate cognition and English language skills to give valid consent and complete research interviews (as assessed by MMSE)
* Willingness to give written informed consent
* Abstinence from alcohol for between 3 and 21 days, and resolution of any clinically evident alcohol withdrawal

Exclusion Criteria:

* Opiate abuse within the last one month
* Sensitivity to study medications or therapy with these drugs within 6 months
* Active major psychiatric disorder associated with psychosis or significant suicide risk
* Pregnancy or lactation
* Advanced decompensated liver disease (hepatocellular failure, variceal bleeding, ascites or encephalopathy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-03; Study Completion 2005-06

PRIMARY OUTCOMES:
Time (days) to relapse
Time (days) to lapse
Days abstinence
Drinks per drinking day
Biochemical measures of liver function

SECONDARY OUTCOMES:
Craving
Depression
Anxiety
Stress
Global physical health
Global mental health

CONTACTS AND LOCATIONS:
Overall Officials: Paul Haber, MBBAMDFRACP, Study Chair — Conjoint Associate Professor
Locations (1):
- Drug Health Services, Royal Prince Alfred Hospital, Sydney, New South Wales, Australia

REFERENCES:
- See also: Click here for more information about this study: The Alcohol Pharmacotherapy Project. This study is run through the University of Sydney. — http://www.alcpharm.med.usyd.edu.au